CLINICAL TRIAL: NCT03008668
Title: Acupuncture for Knee Osteoarthritis With Sensitized Acupoints: a Pilot Randomized Controlled Trial
Brief Title: A Pilot Trial of Acupuncture for Knee Osteoarthritis With Differential Functional Status of Acupoints
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Sun Xin, Director, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201681590955
Record Dates: First submitted 2016-12-26; First posted 2017-01-02 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Acupuncture; Knee Osteoarthritis; Randomized Controlled Trial
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group: Acupuncture (Experimental): acupuncture on 5 most sensitized points/ acupoints
  Interventions: Other: acupuncture
- Control group: Acupuncture (Active Comparator): acupuncture on 5 least low/non-sensitized points
  Interventions: Other: acupuncture

INTERVENTIONS:
Other: acupuncture — a stimulation of the body or auricular points

SUMMARY:
The investigators plan to undertake a rigorous multicentre randomised controlled trial, comparing acupuncture on sensitized acupoints with low/non-sensitive points or no acupuncture (waiting-list), to test if acupuncture on sensitized acupoints may result in improved treatment outcomes in patients with Knee osteoarthritis (KOA).The current pilot study aimed to assess the feasibility of performing the definitive randomised controlled trial.

DETAILED DESCRIPTION:
Patients in the intervention group received acupuncture treatment on the 5 most sensitized points/ acupoints.Patients in the control group received acupuncture treatment on the 5 least /non-sensitized points. All other treatment settings were the same as in the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients are those aged 40 years or older who are diagnosed with KOA and have signed the informed consent.
* The diagnosis of KOA will follow the diagnostic criteria according to the Chinese Guidelines for the Medical Management of Osteoarthritis:
* refractory knee pain for most days in the last month;
* joint space narrowing, sclerosis or cystic change in subchondral bone (as indicated by X-ray);
* laboratory examinations of arthritis: clear and viscous synovial fluid (≥2 times) and white blood cell count < 2000/mm3;
* age 40 years or older;
* morning stiffness continues less than 30 minutes;
* bone sound exists when joints was taking flexion and/or extension. A person is confirmed to be diagnosed with KOA if meeting the either of the three criteria set: (1 and 2), or (1,3 and 5), or (1,4,5 and 6).

Exclusion Criteria:

Patients will be excluded if they:

* Can not adhere to the study protocol in the future 6 months;
* Are diagnosed with conditions leading to skeletal disorders, such as tuberculosis, tumors or rheumatism of knee/bone joint, rheumatoid arthritis;
* Have sprain or other trauma;
* Are unable to walk properly due to foot deformity or pain;
* Are present with mental disorders;
* Have comorbidities including severe cardiovascular disease, liver or kidney impairment, immunodeficiency, diabetes mellitus or blood disorder;
* Females who are pregnant or lactating;
* Were using physiotherapy treatments for osteoarthritis knee pain;
* Had used intra-articular injection of glucocorticoid or viscosupplementation in the past 6 months;
* Received knee-replacement surgery;
* Were participating or had participated in the other clinical trials.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
The change of Western Ontario and McMaster Universities Osteoarthritis index total score from baseline to 16 weeks | Assessments will be conducted at baseline and 16 weeks after randomization
  It consists of 24 items assessing the knee osteoarthritis patients pain, stiffness, and physical function. Each of the 24 items will be graded on a visual analog scale ranging from 0 to 10, with higher scores reflecting more pain, stiffness and poorer physical function

SECONDARY OUTCOMES:
The change of Short Form (SF)-12 health survey score from baseline to 16 weeks | Assessments will be conducted at baseline and 16 weeks after randomization
  It includes 12 items: 2 items on physical functioning, 2 items on role limitations because of physical health problems,
  1 item on bodily pain, 1 item on general health perceptions, 1 item on vitality (energy/fatigue), 1 item on social functioning, 2 items on role limitations because of emotional problems, and 2 items on general mental health (psychological distress and psychological well-being)

OTHER OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Assessments will be conducted at 4 weeks after the acupuncture treatment and followed at 8, 12 and 16 weeks
  Expected adverse events (AEs) of the acupuncture interventions include bleeding, nausea/vomiting, fainting, bruising at needle sites, feeling hot/burning, and transient pain at needle sites. We defined serious adverse events (SAEs) as: death, hospitalization, significant disability or incapacity, any life-threatening situations or any other medically significant events that were potentially related to the trial procedures or acupuncture treatments. The AEs or SAEs were identified by the certified treating acupuncturists.

REFERENCES:
- [Derived] Jia P, Liu J, Li L, Luo Y, Li Y, Zhao L, Liang F, Liu Z, Zou K, Tang L, Sun X. Acupuncture for knee osteoarthritis with sensitized acupoints: results from a pilot, feasibility randomized controlled trial. Pilot Feasibility Stud. 2020 Sep 28;6:144. doi: 10.1186/s40814-020-00687-x. eCollection 2020. PMID 33005432